CLINICAL TRIAL: NCT00517816
Title: A Randomized, Double-blind, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Effect on Pharmacodynamic Biomarkers of an Intravenous Infusion of R1671 in Patients With Mild, Intermittent Asymptomatic Asthma
Brief Title: A Single Ascending Dose Study of R1671 in Patients With Mild Intermittent Asymptomatic Asthma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP21029
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 1 (Experimental)
  Interventions: Drug: RG1671
- 2 (Experimental)
  Interventions: Drug: RG1671
- 3 (Experimental)
  Interventions: Drug: RG1671
- 4 (Experimental)
  Interventions: Drug: RG1671
- 5 (Experimental)
  Interventions: Drug: RG1671
- 6 (Experimental)
  Interventions: Drug: RG1671
- 7 (Experimental)
  Interventions: Drug: RG1671
- 8 (Experimental)
  Interventions: Drug: RG1671

INTERVENTIONS:
Drug: RG1671 — Administered iv at escalating doses (with a starting dose of 0.0015mg)

SUMMARY:
This 8 arm study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of R1671 or placebo in patients with mild, intermittent, asymptomatic asthma. Patients will be randomized to receive placebo or R1671, at a starting dose of 0.0015mg, by intravenous infusion; this dose will be escalated in subsequent groups of patients after a satisfactory assessment of the data from the previous dose. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-50 years of age;
* mild, intermittent, asymptomatic asthma;
* history of asthma for >=6 months;
* non-smokers.

Exclusion Criteria:

* females of childbearing potential, or lactating;
* history of immunologically medicated disease;
* systemic antineoplastic or immunomodulatory treatment in past 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs, ECG. | Throughout study
Serum concentration of R1671, and serum pharmacokinetic parameters. | Throughout study

SECONDARY OUTCOMES:
Pharmacodynamic biomarker sampling; skin prick test. | At intervals during study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Little Rock, Arkansas
  - North Hollywood, California
  - Port Orange, Florida
  - Normal, Illinois
  - Madisonville, Kentucky
  - North Dartmouth, Massachusetts
  - Morrisville, North Carolina
  - San Antonio, Texas